CLINICAL TRIAL: NCT00781092
Title: A Prospective, Randomized, Double-Masked, Single Center, Clinical Comparison of the Use of Systane Ultra in the Management of Dry Eyes in Bilateral Eyes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Durrie Vision (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Principal Investigator, Daniel S. Durrie, MD, President, Durrie Vision
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SUSE-01
Record Dates: First submitted 2008-10-27; First posted 2008-10-28 (Estimated); Last update posted 2012-09-20 (Estimated); Status verified 2012-09

CONDITIONS: Dry Eye
Keywords: Dry Eyes; LASIK; Laser Vision Correction
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Systane Ultra
  Interventions: Other: Systane Ultra
- 2 (Active Comparator): Bausch and Lomb Sensitive Eyes
  Interventions: Other: Bausch and Lomb Sensitive Eyes

INTERVENTIONS:
Other: Systane Ultra — Ophthalmic Solution, 1 gtt, three times daily to both eyes for 1 month post operative
  Other Names: Natural Tears
  Arms: 1
Other: Bausch and Lomb Sensitive Eyes — Ophthalmic Solution, 1 gtt, three times a day in both eyes for 1 month after LASIK
  Other Names: Saline Solution
  Arms: 2

SUMMARY:
The primary objective of this study is to compare two post operative drop regimens for the management of dry eye and control of healing using FDA-approved ophthalmic solutions.

DETAILED DESCRIPTION:
This comparison will be made between bilateral eyes of the same patient following excimer laser ablation using the FDA-approved LADARVision 4000 Excimer Laser System or the WaveLight ALLEGRETTO WAVE™ Excimer Laser System. Post operative questionnaires regarding the use of the drops will be compared. Tear osmolarity and tear breakup time will be evaluated using Tear Lab and OQAS II.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be a suitable candidate for FDA Approved LASIK.
* Subjects must have a stable refraction as documented by previous clinical records.
* Subjects who wear soft contact lenses must discontinue wear at least 3 days prior to preoperative exam or surgery.
* Subjects who wear gas permeable contact lenses must discontinue wear at least 3 weeks prior to preoperative exam or surgery.
* Subjects must be at least 18 years of age.
* Subjects must be willing and able to return for scheduled follow up examinations each day after surgery at the specified time.
* Subjects must sign and be given a copy of the written Informed Consent form.

Exclusion Criteria:

* Subjects for whom either eyes do not meet all inclusion criteria and either eye meets any exclusion criteria.
* Subjects with clinically significant dry eye syndrome or clinically significant blepharitis in either eye.
* Subjects with clinically significant anterior segment pathology, including clinically significant cataracts, corneal scarring or neovascularization in either eye.
* Subjects who have undergone previous intraocular or corneal surgery of any kind, including any type of surgery for either refractive or therapeutic purposes in either eye.
* Subjects who have a history of Herpes zoster or Herpes simplex keratitis.
* Subjects on chronic systemic corticosteroid or other immunosuppressive therapy that may affect wound healing, any immunocompromised subjects, and subjects with clinically significant atopic disease, connective tissue disease, or uncontrolled diabetes.
* Subjects with a history of steroid-responsive rise in intraocular pressure, glaucoma, or preoperative IOP>25 mm Hg in either eye.
* Subjects with macular pathology in either eye.
* Subjects who are pregnant, lactating, or planning to be pregnant during the course of the study.
* Subjects with known sensitivity to planned study concomitant medications.
* Subjects participating in any other ophthalmic drug or device clinical trial during the time of this clinical investigation.
* Use of ocular drugs, other than study medications, during the study and within 30 days prior to study entry or any other ocular medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-10; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Tear osmolarity | 2 week, 1 month

SECONDARY OUTCOMES:
Tear Break Up Time | 2 week, 1 month post op

CONTACTS AND LOCATIONS:
Overall Officials: Daniel S. Durrie, MD, Principal Investigator — Durrie Vision

REFERENCES:
- See also: Durrie Vision Research — http://www.durrievision.com/index.cfm/research